CLINICAL TRIAL: NCT03689244
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Group-sequential, Adaptive, Phase 3 Study With Open-label Extension Period to Assess the Efficacy and Safety of Selexipag as an add-on to Standard of Care Therapy in Subjects With Inoperable or Persistent/Recurrent After Surgical and/or Interventional Treatment Chronic Thromboembolic Pulmonary Hypertension
Brief Title: A Study to Find Out if Selexipag is Effective and Safe in Patients With Chronic Thromboembolic Pulmonary Hypertension When the Disease is Inoperable or Persistent/Recurrent After Surgery and/or Interventional Treatment
Acronym: SELECT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study did not demonstrate efficacy on the primary endpoint, PVR vs. placebo at wk 20 at a planned interim analysis.
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-065B302; 2018-002823-41 (EudraCT Number)
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Results first posted 2023-08-09 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: CTEPH; selexipag
MeSH Terms: interventions — selexipag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Selexipag DB (Experimental): During the double blind treatment period, participants in this group will receive selexipag. Each participant will start with one oral tablet of selexipag 200 µg in the evening of Day 1 and will continue with 200 µg twice daily (b.i.d.) on Day 2. If this dose is well-tolerated, selexipag is up-titrated with weekly increments of 200 µg until reaching the individual maximal tolerated dose (iMTD) in the range of 200 to 1600 µg b.i.d. The up-titration period up to Week 12 is followed by a stable maintenance treatment period from Week 12 to Week 26, at the iMTD. After Week 26, further up-titration can be allowed (but not above 1600 µg b.i.d.).
  Interventions: Drug: Selexipag
- Placebo DB (Placebo Comparator): During the double-blind treatment period, participants in this group will receive the oral matching placebo, twice daily. A (mock) up-titration scheme will be followed.
  Interventions: Drug: Placebo
- Selexipag OL (Experimental): All participants who completed the double-blind treatment period, whether they received placebo or selexipag during the double-blind period, will receive selexipag during the open-label extension period, using the same up-titration schedule as in the double-blind period.
  Interventions: Drug: Selexipag

INTERVENTIONS:
Drug: Selexipag — oral tablets containing 200 µg of selexipag. Depending on the iMTD, participants will receive 1 to 8 tablets at each administration
  Other Names: ACT-293987, JNJ-67896049
  Arms: Selexipag DB; Selexipag OL
Drug: Placebo — Oral tablets without active compound
  Arms: Placebo DB

SUMMARY:
Selexipag is available in many countries for the treatment of pulmonary arterial hypertension (PAH). Due to the similarities between PAH and chronic thromboembolic pulmonary hypertension (CTEPH) and the observed efficacy of other PAH medicines in CTEPH, it is believed that selexipag could benefit to patients with CTEPH. This study aims to assess the efficacy and safety of selexipag in participants with inoperable or persistent/recurrent CTEPH.

DETAILED DESCRIPTION:
Participants will be recruited in two sequential cohorts: approximately the first 90 randomized participants will undergo a right heart catheterization (RHC) (and left heart catheterization LHC, if needed) with measurement of pulmonary vascular resistance (PVR) at Week 20 and will constitute the hemodynamic cohort; the remaining participants will constitute the non-hemodynamic cohort; who do not require a post-baseline hemodynamic assessment. They will undergo the same overall study assessments as the hemodynamic cohort excepted for RHC at Week 20.

ELIGIBILITY:
Main Inclusion Criteria:

* Signed and dated informed consent form
* Male and female participants from greater than or equal to (>) 18 (or the legal age of consent in the jurisdiction in which the study is taking place) and less then or equal to (<=85) years old at Screening (Visit 1)
* With established diagnosis of inoperable CTEPH (i.e., technically non-operable) or persistent/recurrent CTEPH after pulmonary endarterectomy (PEA) and/or balloon pulmonary angioplasty (BPA), as confirmed by the corresponding adjudication committee
* With pulmonary hypertension (PH) in WHO FC I-IV.
* Participant able to perform the 6-minute walk test (6MWT) with a minimum distance of 100 m and a maximum distance of 450 m at screening visit.
* Women of childbearing potential must have a negative pregnancy test at screening and randomization and must agree to undertake monthly urine pregnancy tests, and to use a reliable method of birth control from screening visit up to at least 30 days after study treatment discontinuation. If a hormonal contraceptive is chosen it must be taken for at least 1 month prior to randomization.

Main Exclusion Criteria:

* Planned or current treatment with another investigational treatment up to 3 months prior to randomization.
* Any known factor or disease that might interfere with treatment compliance, study conduct, or interpretation of the results, such as drug or alcohol dependence or psychiatric disease.
* Known concomitant life-threatening disease with a life expectancy < 12 months.
* Planned balloon pulmonary angioplasty within 26 weeks after randomization.
* Change in dose or initiation of new PH-specific therapy within 90 days prior to the baseline RHC (and LHC, if needed) qualifying for enrollment for the hemodynamic cohort and within 90 days prior to randomization (Visit 2) for the non-hemodynamic cohort
* Treatment with prostacyclin (epoprostenol), prostacyclin analogs (i.e., treprostinil, iloprost, beraprost) or prostacyclin receptor agonists (i.e., selexipag) within 90 days prior to randomization (visit 2) except those given at vasodilator testing during RHC
* Change in dose or initiation of new diuretics and/or calcium channel blockers within 1 week prior to baseline RHC (and LHC, if needed)
* Any co-morbid condition that may influence the ability to perform a reliable and reproducible 6MWT, including use of walking aids (cane, walker, etc).
* Any other criteria as per selexipag Summary of Product Characteristics (SmPC).
* Exclusion criteria related to comorbidities: severe coronary heart disease or unstable angina as assessed by the investigator; mocardial infarction within the last 6 months prior to or during Screening; decompensated cardiac failure if not under close supervision; severe arrhythmias as assessed by the investigator; cerebrovascular events (example transient ischemic attack, stroke) within the last 3 months prior to or during screening; congenital or acquired valvular defects with clinically relevant myocardial function disorders not related to pulmonary hypertension. (PH); known or suspicion of pulmonary veno-occlusive disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Borissoff, MD, PhD, Study Director — Actelion
Locations (162):
- United States (32):
  - University of California San Diego Medical Center, La Jolla, California
  - University of Southern California, Keck School of Medicine, Los Angeles, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Colorado Springs Pulmonary Consultants, Colorado Springs, Colorado
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago Hospitals - Chicago, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Maryland, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - St. Mary's Cardiology, Reno, Nevada
  - University of New Mexico Clinical & Translational Science Center, Albuquerque, New Mexico
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Baylor Scott & White Research Institute at The Heart Hospital Baylor Plano, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Cardiovascular Center, Salt Lake City, Utah
  - Medical College of Wisconsin Froedtert Hospital, Milwaukee, Wisconsin
  - Aurora Saint Lukes Medical Center, Milwaukee, Wisconsin
- Argentina (7):
  - Sanatorio de la Trinidad Mitre, Buenos Aires
  - Centro Médico Dra. De Salvo, Buenos Aires
  - Hospital Italiano de Buenos Aires, Caba
  - Sanatorio Ramon Cereijo, Caba
  - Instituto de Cardiología y Cirugía Cardiovascular - Fundación Favaloro, Caba
  - Hospital General de Agudos Dr Cosme Argerich, CABA
  - Hospital Britanico de Buenos Aires, CABA
- Australia (6):
  - Royal Adelaide Hospital, Adelaide
  - Queensland Lung Transplant Service, Chermside
  - St Vincent's hospital, Darlinghurst
  - Pulmonary Arterial Hypertension Clinic, Hobart
  - The Alfred Hospital, Melbourne
  - Westmead Hospital, Westmead
- Austria (2):
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Medical University Vienna, Vienna
- Belgium (2):
  - ULB Hôpital Erasme, Brussels
  - UZ Leuven, Leuven
- Brazil (11):
  - Universidade Federal De Minas Gerais - Hospital das Clínicas, Belo Horizonte
  - Instituto das Pequenas Missionárias de Maria Imaculada - Hospital Madre Teresa, Belo Horizonte
  - Fundacao para o Desenvolvimento Medico Hospitalar (UNESP Botucatu), Botucatu
  - Secretaria da Saude do Estado do Ceara - Hospital Doutor Carlos Alberto Studart Gomes, Fortaleza
  - Universidade Federal de Goias - Hospital das Clinicas da UFG, Goiânia
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre
  - Fundacao do ABC - Centro Universitario FMABC, Santo André
  - SPDM - Associacao Paulista para o Desenvolvimento da Medicina - Hospital Sao Paulo, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- Bulgaria (3):
  - UMHAT 'Heart and Brain Center for Excellence', Pleven
  - National Cardiology Hospital, Sofia
  - University Multiprofile Hospital for Active Treatment- UMHAT Sveta Anna AD, Sofia
- Canada (5):
  - University Of Calgary - Peter Lougheed Centre, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Institut Universitaire De Cardiologie Et De Pneumologie De Québec, Québec, Quebec
- China (6):
  - Chinese Academy of Medical Sciences(CAMS) & Peking Union Medical College(PUMC), Beijing
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The General Hospital of Northern Theater Command, Shenyang
  - Shengjing Hospital Of China Medical University, Shenyang
  - Shanxi Cardiovascular Hospital, Taiyuan
  - Tianjin Medical University General Hospital, Tianjin
- General University Hospital II.department of Internal Medicine-cardiology and angiology, Prague, Czechia
- Denmark (2):
  - Århus Universitetshospital, Skejby, Hjertemedicinsk Afdeling B, Aarhus
  - Rigshospitalet Kardiologisk Klinisk, Copenhagen
- Germany (9):
  - Universitätsklinikum Carl Gustav Carus Medizinische Klinik und Poliklinik 1-Pneumologie, Dresden
  - Universitätsklinikum Giessen Medizinische Klinik Und Poliklinik Ii, Pneumologie, Giessen
  - Universität Greifswald - Klinik Für Innere Medizin Bereich Pneumologie/Infektiologie, Greifswald
  - Universitätsklinikum Hamburg-Eppendorf - Pneumologie, Hamburg
  - Medizinische Hochschule Hannover Zentrum Innere Medizin Klinik für Pneumologie, Hanover
  - Thoraxklinik am Universitatsklinikum Heidelberg, Heidelberg
  - Universitätskliniken des Saarlandes / Medizinische Klinik und Poliklinik, Innere Medizin V, Homburg/Saar
  - Universitätsklinikum Leipzig Medizinischen Klinik und Poliklinik I, Abteilung für Pneumologie, Leipzig
  - Klinikum Würzburg Mitte gGmbH Standort Missioklinik, Würzburg
- Hungary (5):
  - Semmelweis Egyetem,Pulmonológiai Klinika, Budapest
  - Gottsegen György Országos Kardiológiai Intézet, Felnőtt kardiológiai osztály, Budapest
  - Debreceni Egyetem Orvos es Egeszsegtudomanyi Centrum, Debrecen
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Szegedi Tudományegyetem, Általános Orvostudományi Kar, Családorvosi Intézet és rendelő, Szeged
- Israel (2):
  - Rabin Medical Center Beilinson Campus, Petah Tikva
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (4):
  - Azienda Ospedaliera Policlinico S. Orsola-Malpighi, Bologna
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Policlinico Umberto I, Roma
  - Ospedale di Cattinara - Struttura complessa di Pneumologia, Trieste
- Malaysia (3):
  - Hospital Pulau Pinang, George Town
  - Hospital Serdang, Kajang
  - Institut Jantung Negara (National Heart Institute), Kuala Lumpur
- Mexico (3):
  - CICUM San Miguel, Guadalajara
  - Instituto Nacional de Cardiologia Dr. Ignacio Chavez, Mexico City
  - Unidad de Investigacion Clinica en Medicina S.C. (UDICEM), Monterrey
- Netherlands (2):
  - VUMC Amsterdam, Amsterdam
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
- Poland (8):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Krakowski Szpital Specjalistyczny im Jana Pawla II, Krakow
  - Wojewodzki Szpital Specjalistyczny im. Stefana Kardynala Wyszynskiego SPZOZ, Lublin
  - NZOZ Europejskie Centrum Zdrowia Otwock, Otwock
  - Uniwersytet Medyczny im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Samodzielny Publiczny Szpital Kliniczny nr 2 PUM, Szczecin
  - Warszawski Uniwersytet Medyczny, Szpital Kliniczny Dzieciątka Jezus, Warsaw
  - Wojewodzki Szpital Specjalist, Osrodek Badawczo-Rozwojowy, Wroclaw
- Portugal (4):
  - Hospital Garcia de Orta, Almada
  - Hospitais da universidade de Coimbra, Coimbra
  - Centro Hospitalar de Lisboa Norte, Lisbon
  - Hospital Geral de Santo Antonio, Porto
- Russia (7):
  - Irkutsk Regional Clinical Hospital, Irkutsk
  - Cardiovascular Pathology Research Institute of Siberian Branch of RAMS, Kemerovo
  - Moscow City Clinical Hospital #1 n.a. N.I.Pirogov, Moscow
  - Moscow City Clinical Hospital No.51, Moscow
  - National Medical Research Center of Cardiology of MoH of Russian Federation, Moscow
  - E.Meshalkin National Medical Research Center of the Ministry of Health of the Russian Federation, Novosibirsk
  - National medical Research Center n.a. V.A.Almazov of MoH of Russian Federation, Saint Petersburg
- Narodny ustav srdcovych a cievnych chorob, Bratislava, Slovakia
- South Korea (5):
  - Pusan National University Hospital, Busan
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (6):
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. Vall D Hebron, Barcelona
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Univ. I Politecni La Fe, Valencia
- Sweden (2):
  - Norrlands Universitetssjukhus, Umeå
  - Uppsala Akademiska Sjukhuset, Kardiologkliniken, Uppsala
- Universitatsspital Zurich, Zurich, Switzerland
- Taiwan (4):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Thailand (2):
  - Ramathibodi Hospital Mahidol University, Bangkok
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
- Turkey (Türkiye) (7):
  - Hacettepe University Medical Faculty, Ankara
  - Ankara University Medical Faculty, Ankara
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Marmara University Medical Faculty, Istanbul
  - Ege University Medical Faculty, Izmir
  - Kartal Kosuyolu Yuksek Ihtisas Egitim Ve Arastirma Hastanesi, Kartal Istanbul
- Ukraine (4):
  - CE 'Dnipropetrovsk Regional Clinical Center of Cardiology and Cardiosurgery', Dnipro
  - SI National Scientific Center Institute of Cardiology of M.D. Strazhesko of NAMS of Ukraine, Kyiv
  - SI 'National Institute of Phtisiology and Pulmonology n.a. F.G. Yanovsky of NAMS of Ukraine', Kyiv
  - Lviv Regional Clinical Hospital, Lviv
- United Kingdom (6):
  - Papworth Hospital NHS Trust, Cambridge
  - National Waiting Times Centre Board Golden Jubilee National Hospital, Glasgow
  - Royal Free Hospital, London
  - Royal Brompton Hospital, London
  - Hammersmith Hospital, London
  - Sheffield Teaching Hospitals NHS Foundation Trust Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Actelion is a Janssen pharmaceutical company of Johnson & Johnson. The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials\transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Kim NH, Channick R, Delcroix M, Madani M, Pepke-Zaba J, Borissoff JI, Easton V, Gesang S, Richard D, Ghofrani HA. Efficacy and safety of selexipag in patients with inoperable or persistent/recurrent CTEPH (SELECT randomised trial). Eur Respir J. 2024 Oct 3;64(4):2400193. doi: 10.1183/13993003.00193-2024. Print 2024 Oct. PMID 39326918

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 321 participants were screened, of which 128 were randomly assigned and received study intervention.
Groups:
- Double-blind Period: Placebo: Participants received a single oral tablet of placebo matching to selexipag 200 micrograms (mcg) in the evening of Day 1 and continued the same dose (200 mcg) twice daily (BID) on Day 2. Upon first dose toleration, placebo dose was up-titrated with weekly increments of 200 mcg until reaching the individual maximum tolerated dose (iMTD) in the range of 200 to 1600 mcg BID. The up-titration up to Week 12 was followed by a stable maintenance treatment period with the iMTD (reached at Week 12) until Week 26. After Week 26 up to end of DB treatment (EDBT) period, further up-titration was done but not above 1600 mcg, BID (maximum duration: 24.6 months). For participants with moderate hepatic impairment (Child-Pugh B) or who were concomitantly taking a moderate Cytochrome P-450 2C8 (CYP2C8) inhibitor, the dosing frequency was to be once daily (QD).
- Double-blind Period: Selexipag: Participants received a single oral tablet of selexipag 200 mcg in the evening of Day 1 and continued the same dose (200 mcg) BID on Day 2. Upon first dose toleration, selexipag dose was up-titrated with weekly increments of 200 mcg until reaching the iMTD in the range of 200 to 1600 mcg BID. The up-titration up to Week 12 was followed by a stable maintenance treatment period with the iMTD (reached at Week 12) until Week 26. After Week 26 up to EDBT period, further up-titration was done but not above 1600 mcg, BID (maximum duration: 27.7 months). For participants with moderate hepatic impairment (Child-Pugh B) or who were concomitantly taking a moderate CYP2C8 inhibitor, the dosing frequency was to be QD.
- Open Label Period: Selexipag (Ex-Placebo): All participants (received placebo in DB period) who completed DB treatment period, entered OL extension period and received the first dose (selexipag 200 mcg) of OL period in the evening of the EDBT and then selexipag 200 mcg BID on the day after. Participants with moderate hepatic impairment (Child-Pugh B) or who had taken concomitantly moderate CYP2C8 inhibitor(s) started one tablet of OL selexipag 200 mcg in the morning of the day after EDBT visit. Dose up-titration was done as like DB treatment till iMTD was reached. The up-titration up to Week 12 was followed by a stable maintenance treatment period with the iMTD (reached at Week 12) until Week 26. After Week 26 up to end of OL treatment (EOLT) period, further up-titration was done but not above 1600 mcg, BID (maximum duration: 20.8 months).
- Open Label Period: Selexipag (Ex-Selexipag): All participants (received selexipag in DB period) who completed DB treatment period, entered OL extension period and received the first dose (selexipag 200 mcg) of OL period in the evening of the EDBT and then selexipag 200 mcg BID on the day after. Participants with moderate hepatic impairment (Child-Pugh B) or who had taken concomitantly moderate CYP2C8 inhibitor(s) started one tablet of OL selexipag 200 mcg in the morning of the day after EDBT visit. Dose up-titration was done as like DB treatment till iMTD was reached. The up-titration up to Week 12 was followed by a stable maintenance treatment period with the iMTD (reached at Week 12) until Week 26. After Week 26 up to EOLT period, further up-titration was done but not above 1600 mcg, BID (maximum duration: 19.8 months).
Period: Double Blind Period (Up to 27.7 Months)
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Selexipag | Open Label Period: Selexipag (Ex-Placebo) | Open Label Period: Selexipag (Ex-Selexipag)
Started | 64 | 64 | 0 | 0
Completed | 9 | 6 | 0 | 0
Not Completed | 55 | 58 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 8 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0
Not completed — Sponsor decision | 44 | 47 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 2 | 0 | 0
Period: Open Label Period (Up to 20.8 Months)
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Selexipag | Open Label Period: Selexipag (Ex-Placebo) | Open Label Period: Selexipag (Ex-Selexipag)
Started | 0 | 0 | 9 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 9 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Sponsor Decision | 0 | 0 | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Selexipag | Total
Number analyzed (Participants) | 64 | 64 | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 36 | 60
  >=65 years | 40 | 28 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (13.22) | 62 (14.38) | 63 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 46 | 93
  Male | 17 | 18 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 18
  Not Hispanic or Latino | 54 | 55 | 109
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 12 | 7 | 19
  Black or African American | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 46 | 52 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
  Other | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 0 | 2 | 2
  AUSTRALIA | 1 | 3 | 4
  BELGIUM | 0 | 1 | 1
  BRAZIL | 5 | 6 | 11
  BULGARIA | 1 | 3 | 4
  CANADA | 0 | 1 | 1
  CHINA | 0 | 2 | 2
  CZECH REPUBLIC | 1 | 2 | 3
  DENMARK | 4 | 3 | 7
  GERMANY | 6 | 9 | 15
  HUNGARY | 0 | 1 | 1
  ISRAEL | 2 | 0 | 2
  ITALY | 2 | 3 | 5
  MEXICO | 4 | 1 | 5
  POLAND | 2 | 2 | 4
  PORTUGAL | 5 | 1 | 6
  RUSSIAN FEDERATION | 4 | 3 | 7
  SLOVAKIA | 0 | 1 | 1
  SOUTH KOREA | 7 | 2 | 9
  SPAIN | 1 | 0 | 1
  SWEDEN | 0 | 1 | 1
  TAIWAN | 1 | 1 | 2
  THAILAND | 4 | 2 | 6
  TURKEY | 4 | 4 | 8
  UKRAINE | 0 | 1 | 1
  UNITED KINGDOM | 5 | 6 | 11
  UNITED STATES | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pulmonary Vascular Resistance (PVR) at Week 20
Description: Change from baseline in PVR at Week 20 was reported. PVR was measured by accessing the vessel either from right heart catheterization or left heart catheterization, if required. Change from baseline in PVR was measured as percent ratio of post treatment value (Week 20) to pre-treatment value (baseline).
Time Frame: Baseline (Day 1, pre-dose), within 2 to 5 hours post-dose on Week 20
Population: Hemodynamic set (HES) included all assigned participants in the hemodynamic cohort.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Percent ratio
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Selexipag
Number analyzed (Participants) | 44 | 47
Percent ratio | 89.52 [81.78 to 97.99] | 85.15 [77.97 to 92.99]
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Selexipag; Ratio of Geometric mean of Selexipag to Placebo was reported; Test type: Superiority; p = 0.412, ANCOVA; Ratio of Geometric LS mean = 0.95, 95% CI 2-sided [0.84 to 1.07]

ADVERSE EVENTS:
Time Frame: For DB period: from first DB dose up to EDBT (that is, up to 27.7 months) and for OL extension period: from first OL dose up to 30 days after the last OL dose (that is, up to 21.8 months)
Description: Safety analysis set (SAF) included all participants who received at least one dose of study treatment.
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Selexipag | Open Label Period: Selexipag (Ex-Placebo) | Open Label Period: Selexipag (Ex-Selexipag)
All-Cause Mortality (participants affected / at risk) | 2/64 | 3/64 | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 16/64 | 9/64 | 0/9 | 1/6
Other Adverse Events (participants affected / at risk) | 45/64 | 60/64 | 9/9 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Period: Placebo (N=64) | Double-blind Period: Selexipag (N=64) | Open Label Period: Selexipag (Ex-Placebo) (N=9) | Open Label Period: Selexipag (Ex-Selexipag) (N=6)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrial Flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 0 | 0 | 0
Right Ventricular Failure (Cardiac disorders) | 3 | 5 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Discoloured Vomit (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Catheter Site Haematoma (General disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 1 | 0 | 0
Hepatitis Acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Covid-19 Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia Bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Septic Shock (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Urethral Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 1 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Period: Placebo (N=64) | Double-blind Period: Selexipag (N=64) | Open Label Period: Selexipag (Ex-Placebo) (N=9) | Open Label Period: Selexipag (Ex-Selexipag) (N=6)
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 1 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 6 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 4 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 5 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 38 | 5 | 1
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 17 | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 11 | 3 | 1
Asthenia (General disorders) | 0 | 3 | 1 | 0
Chest Pain (General disorders) | 3 | 2 | 1 | 0
Fatigue (General disorders) | 4 | 6 | 0 | 0
Oedema (General disorders) | 3 | 0 | 1 | 0
Oedema Peripheral (General disorders) | 8 | 5 | 0 | 0
Pain (General disorders) | 0 | 5 | 0 | 1
Covid-19 (Infections and infestations) | 4 | 5 | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Blood Glucose Increased (Investigations) | 0 | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 6 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Steroid Diabetes (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 14 | 3 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 7 | 4 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 13 | 1 | 1
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 2 | 16 | 2 | 0
Dizziness (Nervous system disorders) | 7 | 8 | 2 | 0
Headache (Nervous system disorders) | 14 | 36 | 6 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 0 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1
Flushing (Vascular disorders) | 2 | 4 | 1 | 1
Hot Flush (Vascular disorders) | 0 | 2 | 0 | 1
Hypotension (Vascular disorders) | 4 | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
Failure to meet success on the primary outcome measure led to termination of the study for futility and thus the pre-planned testing hierarchy was no longer applicable, and all efficacy analyses other than the primary endpoint (PVR) were exploratory.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 30 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filling of a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/44/NCT03689244/Prot_002.pdf
  • Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT03689244/SAP_003.pdf